CLINICAL TRIAL: NCT01819467
Title: A Randomized Controlled Trial to Reduce Adhesions Following a Primary Cesarean Section
Brief Title: A Trial to Reduce Adhesions Following a Primary Cesarean Section
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow to accrue, lack of qualified participants
Sponsor: South East Area Health Education Center, Wilmington, NC (Other)
Collaborators: New Hanover Regional Medical Center (Other)
Responsible Party: Principal Investigator, Todd Beste, Chair/Program Director of Residency Program Department of Obstetrics & Gynecology NH NHRMC, South East Area Health Education Center, Wilmington, NC
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1301-1
Record Dates: First submitted 2013-03-18; First posted 2013-03-27 (Estimated); Results first posted 2023-08-16 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-07

CONDITIONS: Tissue Adhesions
MeSH Terms: conditions — Tissue Adhesions

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Group (Active Comparator): Patients in this group will receive Seprafilm onto the uterine incision and the anterior midline of the uterus.
  Interventions: Device: Seprafilm
- Control Group (No Intervention): This arm will be known as the control/no intervention group. This group will not receive Seprafilm or any other adhesion barrier method

INTERVENTIONS:
Device: Seprafilm — Seprafilm will be placed onto the uterine incision and the anterior midline of the uterus following the primary cesarean section
  Arms: Treatment Group

SUMMARY:
The primary objective of this study is to determine whether the use of Seprafilm reduces the incidence rate of adhesion formation following a primary C-section.

A secondary objective of the study will be to determine whether or not a correlation between the adhesion score and the difficulty or delay in delivery of the infant exists.

DETAILED DESCRIPTION:
A cesarean section or delivery (C-section/CD) is the surgical removal of an infant and placenta through the mother's abdominal and uterine wall. This procedure is performed by an obstetrician and is one of the most common types of surgical methods used today. According to the Centers for Disease Control and Prevention, the rate for this method of delivery has risen over the past decade. However, recent research has shown that patients who receive this surgical procedure become more susceptible to adhesions.

Adhesions are formations (bands) of scar tissue that occur immediately following most surgical procedures. Adhesions limit the mobility of tissues and organs near the incision site by causing them to stick together. This limited mobility can generate an increased rate of morbidity (occurrence of other diseases). Morbidities caused by adhesions include but are not limited to abdominal and/or pelvic pain, bowel obstruction (partial or complete blockage of the bowel), subfertility (difficulty getting pregnant) and infertility (inability to get pregnant).

A study conducted by Dierdre Lyell, MD reported that the incidence of adhesion formation following a primary CD ranges from 46-65%. Another study (Morales et al) reported that for women who had undergone a CD, the incidence rate of adhesions and severe adhesions was greater in women who had had repeat CDs compared with women who only had a primary CD. In addition, this study also states that the percentage of adhesion occurrence increases in women with each subsequent (following) CD.

Numerous methods have been implemented toward the preventions of adhesions. Currently, Seprafilm is an approved adhesion prevention method that is used in most surgical procedures. Seprafilm is a clear film that is composed of chemically modified sugars (some of which occur naturally in the human body). Unlike its counterpart Interceed, Seprafilm is unaffected by the presence of blood. After being placed, Seprafilm becomes a gel within 24-48 hours and then is slowly absorbed and excreted by the body over the course of 1-4 weeks.

Seprafilm Adhesion Barrier is FDA approved for use in patients undergoing abdominal or pelvis laparotomy as an adjunct intended to reduce the incidence, extent and severity of post-operative adhesions between the abdominal and between the uterus and surrounding structures.

ELIGIBILITY:
Inclusion Criteria:

* Females 12 years and older undergoing a scheduled primary cesarean section at or after 24 weeks estimated gestational period

Exclusion Criteria:

* Patients transferred from outlying hospitals who expect to undergo repeat C-section at that hospital.
* Patients who have had previous laparotomy
* Patients having a previous laparoscopy demonstrating adhesions of bladder peritoneum or uterine serosa or myometrium to the parietal peritoneum or omentum or bowel to the uterus or parietal peritoneum; or involving pelvic adhesiolysis, enterolysis or other surgery on bowel located in the pelvis, uterine myomectomy , adnexectomy or other adnexal surgery including ovarian cystectomy, tuboplasty, tubal reanastomosis, and removal of endometriosis
* Patients with an adhesion score > 0 at the time of primary cesarean section
* Patents with chorioamnionitis, appendicitis or infection of other pelvic viscera at the time of primary cesarean section.
* Patients who have taken systemic corticosteroids within 2 weeks of the primary cesarean section. Provided however, patients who have been treated with systemic betamethasone or dexamethasone to promote fetal lung maturity are not excluded
* Patients undergoing tubal sterilization at the time of the primary cesarean section
* Patients with known allergy to hyaluronic acid
* The following criteria are seen as complications or adverse events experienced by the patients in the interval after the puerperium and will therefore exclude patients:

  1. Patient who have had a pelvic inflammatory disease documented by either cervical motion, uterine or adnexal tenderness; and either oral temperature > 101 degrees or mucopurulent cervical discharge or cervical culture positive for C. trachomatis or N. Gonorrhoeae
  2. Patients who have pelvic abscess or diverticulitis

Min Age: 12 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry A Easley, MD, Principal Investigator — South East Area Health Education Center
Locations (1):
- New Hanover Regional Medical Center, Wilmington, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Morales KJ, Gordon MC, Bates GW Jr. Postcesarean delivery adhesions associated with delayed delivery of infant. Am J Obstet Gynecol. 2007 May;196(5):461.e1-6. doi: 10.1016/j.ajog.2006.12.017. PMID 17466702
- [Background] Lyell DJ. Adhesions and perioperative complications of repeat cesarean delivery. Am J Obstet Gynecol. 2011 Dec;205(6 Suppl):S11-8. doi: 10.1016/j.ajog.2011.09.029. Epub 2011 Oct 6. PMID 22114993

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Scheduled C-section deliveries
Pre-assignment Details: Non-C-section deliveries
Groups:
- Seprafilm: Patients in this group will receive Seprafilm onto the uterine incision and the anterior midline of the uterus.
  Seprafilm: Seprafilm will be placed onto the uterine incision and the anterior midline of the uterus following the primary cesarean section
- Control: No Seprafilm was placed on to the uterine incision.
Period: Overall Study
Arm/Group | Seprafilm | Control
Started (29) | 20 | 9
Completed (Study terminated) | 0 | 0
Not Completed | 20 | 9
Not completed — Physician Decision | 20 | 9

BASELINE CHARACTERISTICS:
Population: Pregnant females ages 12 and older
Groups:
- Seprafilm: Pregnant females age 12 and over who underwent a C-Section and Seprafilm was placed on the uterine incision.
- Control: Did not receive Seprafilm on uterine incision.
- Total: Total of all reporting groups
Arm/Group | Seprafilm | Control | Total
Number analyzed (Participants) | 20 | 9 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 9 | 29
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Female
  Participants
    Female | 20 | 9 | 29
    Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Adhesion Formation Following a Primary C-section With and Without Adhesion Barrier
Description: Study was terminated due to too many protocol deviations. There were no outcome measures analyzed.
Time Frame: 21 months
Population: No data for pre-specified Primary and Secondary Outcome Measures were collected.
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 21 months
Groups:
- Seprafilm Group: This group received seprafilm.
- Control Group: This group will not receive seprafilm
Arm/Group | Seprafilm Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/9
Other Adverse Events (participants affected / at risk) | 0/20 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes